CLINICAL TRIAL: NCT04430140
Title: CT Scalar Localization of the Electrode Array Following Cochlear Implantation
Brief Title: CT Scalar Localization
Status: Withdrawn | Type: Observational
Why Stopped: Alternative study opened with ENT services.
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, John Lane, Principal Investigator, Mayo Clinic
Other Study IDs: 19-005543
Record Dates: First submitted 2020-06-08; First posted 2020-06-12 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Cochlear Implant
MeSH Terms: interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: CT Scan
  Number of research exams: 1 Effective Dose (mSv) for 1 exam: 0.6 Total Effective Dose (mSv)*: 0.6
  Interventions: Device: CT Scan

INTERVENTIONS:
Device: CT Scan — CT Scan
  Number of research exams: 1 Effective Dose (mSv) for 1 exam: 0.6 Total Effective Dose (mSv)*: 0.6

SUMMARY:
Comparing the location of cochlear implants to level of retained hearing.

DETAILED DESCRIPTION:
Subjects who have undergone cochlear implant surgery will have a CT scan to determine the exact anatomical location of the implant. This location will then be compared with audio testing levels and operative reports to determine any advances in implantation technique that would result in more preserved hearing

ELIGIBILITY:
Inclusion Criteria:

* Currently scheduled for a cochlear implant or currently have a cochlear implant
* 18 years of age and over
* Male and female
* Capacity to consent for patients will be determined by review of the medical history of subject at screening and in concert with the referring physician. Consent will be signed after all questions have been answered and the participant indicates they understand

Exclusion Criteria:

* Younger than 18 years of age
* Current criteria for cochlear implantation
* Currently pregnant, all females will be asked to take a urine pregnancy test if of child bearing age, unless you cannot become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mayo Clinic Patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Implant Location | 3 Years
  Determining location of implant using CT scan and correlating retained hearing levels

CONTACTS AND LOCATIONS:
Overall Officials: John Lane, MD, Principal Investigator — Mayo Clinic

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials